CLINICAL TRIAL: NCT02813967
Title: S-1 Concurrent With Radiotherapy Versus Radiotherapy for Elderly Chinese Patients With Squamous Cell Carcinoma of Esophagus: A Prospective, Randomized, Multi-center Phase-III Study
Brief Title: S-1 Concurrent With Radiotherapy Versus Radiotherapy for Elderly Patients With Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-E-E
Record Dates: First submitted 2016-06-14; First posted 2016-06-27 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Esophageal Cancer; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemoradiotherapy (Experimental): Radiotherapy 54 Gy was administered in 1.8 Gy fractions 5 times weekly. S-1 70mg/m2 was administered on days 1-14 and 29-42
  Interventions: Radiation: Radiotherapy 54 Gy; Drug: S-1
- Radiotherapy 60 Gy (Active Comparator): Radiotherapy 60 Gy was administered in 2Gy fractions 5 times weekly.
  Interventions: Radiation: Radiotherapy 60 Gy

INTERVENTIONS:
Radiation: Radiotherapy 54 Gy — Radiotherapy was administered in 1.8 Gy fractions 5 times weekly to a total dose of 54 Gy.
  Arms: chemoradiotherapy
Radiation: Radiotherapy 60 Gy — Radiotherapy was administered in 2 Gy fractions 5 times weekly to a total dose of 60Gy.
  Arms: Radiotherapy 60 Gy
Drug: S-1 — S-1 70mg/m2 was administered on days 1-14 and 29-42.
  Arms: chemoradiotherapy

SUMMARY:
This was a randomised, multicenter, phase 3 trial. Patients who were age of 70 years or older with histologically confirmed esophageal cancer were randomly assigned to S-1 concurrent with radiotherapy or radiotherapy alone.The primary endpoint was overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic diagnosis of esophageal carcinoma
* ECOG performance status 0-1
* Age:70-85 years
* Joined the study voluntarily and signed informed consent form
* Patients must not have received any prior anticancer therapy
* Stage Ⅰ-ⅣB（AJCC 2009）
* Target lesions can be measured according to RECIST criteria
* No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥9 g/dL, WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L, platelet count ≥100x 109/L, TBIL<1.5 x ULN, ALT and AST ≦ 2.5 x ULN, creatinine ≦ 1.5 x ULN

Exclusion Criteria:

* Multiple carcinomas of the esophagus,
* Biopsy-proven invasion of the tracheobronchial tree or tracheoesophageal fistula,
* Metastatic disease (M1b),
* A primary tumor that extended to within 2 cm of the gastroesophageal junction,
* Prior chemotherapy, prior thoracic radiation, surgical resection of the primary tumor,
* history of a second malignancy other than nonmelanoma skin cancer

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-06; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  2-year over survival

SECONDARY OUTCOMES:
Progression-free survival | 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years

OTHER OUTCOMES:
the quality of life | 5 years
  assessed with the European Organisation for Research and Treatment of Cancer quality-of-life core questionnaire QLQ-C30
the oesophagus-specific quality-of-life | 5 years
  assessed with the European Organisation for Research and Treatment of Cancer quality-of-life the oesophagus-specific questionnaire QLQ-OES18

CONTACTS AND LOCATIONS:
Overall Officials: MING CHEN, PHD, Study Chair — Zhejiang Cancer Hospital; XIANGHUI DU, MD, Principal Investigator — Zhejiang Cancer Hospital; youngling JI, MD, Study Director — Zhejiang Cancer Hospital; weiguo zhu, MD, Study Director — Huaian first people's hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji Y, Du X, Zhu W, Yang Y, Ma J, Zhang L, Li J, Tao H, Xia J, Yang H, Huang J, Bao Y, Du D, Liu D, Wang X, Li C, Yang X, Zeng M, Liu Z, Zheng W, Pu J, Chen J, Hu W, Li P, Wang J, Xu Y, Zheng X, Chen J, Wang W, Tao G, Cai J, Zhao J, Zhu J, Jiang M, Yan Y, Xu G, Bu S, Song B, Xie K, Huang S, Zheng Y, Sheng L, Lai X, Chen Y, Cheng L, Hu X, Ji W, Fang M, Kong Y, Yu X, Li H, Li R, Shi L, Shen W, Zhu C, Lv J, Huang R, He H, Chen M. Efficacy of Concurrent Chemoradiotherapy With S-1 vs Radiotherapy Alone for Older Patients With Esophageal Cancer: A Multicenter Randomized Phase 3 Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1459-1466. doi: 10.1001/jamaoncol.2021.2705. PMID 34351356